CLINICAL TRIAL: NCT03542227
Title: Study for the Development of Standard Operating Procedures for Anti-HPV Antibody Detection in First-void Urine: the AB-SOP Follow-up Study
Brief Title: Standard Operating Procedures for Anti-HPV (Human Papillomavirus) Antibody Detection in First-void Urine
Acronym: ABSOP-FollowUp
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, Principal investigator, Universiteit Antwerpen
Other Study IDs: B300201734258
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Human Papilloma Virus Infection
Keywords: Antibodies; Vaccination; Self-sampling; First-void urine; HPV
MeSH Terms: conditions — Papillomavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First-void urine samples (3) and serum samples (1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: First-void urine collection — Collection of ca. 20 ml of first-void urine with the Colli-PeeTM device (Novosanis) during visit at the Centre for the Evaluation of Vaccination.
  Other Names: FV urine
Other: Blood draw — Blood sample collection (5-10 cc) by a study nurse of Centre for the Evaluation of Vaccination.
  Other Names: Serum sample

SUMMARY:
The aim of the study is to develop and implement robust analytical protocols for first-void urine sample preparation and antibody assays to monitor vaccine induced immunity against HPV (Human Papillomavirus).

DETAILED DESCRIPTION:
Participants of the HPV V503-004 study (Phase III Clinical trial vaccinating (young) adult women in Antwerp, EudraCT NUMBER: 2015-005093-38) will be asked if they are willing to provide two additional urine samples at day 1 and month 7 for biomedical research. Furthermore, they will be contacted again at approximately 3.5 years and asked if they are willing to provide an additional urine sample and a serum sample. At 3.5 years, they will also be asked to fill in a brief questionnaire. The collected urine will be used for the development and optimization of robust analytical protocols for sample preparation and antibody assays.

ELIGIBILITY:
Inclusion Criteria:

* Participant of the HPV V503-004 study at UA/UZA
* Willing to give informed consent (ICF) to the CEV research team

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In total 63 women are included in this trial. During their first two study visits, at day 0 and 7m post-vaccination, participants are asked to collect a first-void urine sample with the Colli-PeeTM device (n=63). During their third visit, the included women are asked to collect a third first-void urine sample with the Colli-PeeTM device (n = 58). Hereafter, a blood sample of 5-10 cc is collected. Following sample collection, women are asked to fill in a questionnaire (n=58).
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Concentration of HPV specific IgG (Immunoglobulin G) in FV urine. | Within 6 months after study completion
  To detect HPV specific IgG concentrations (ratio HPV specific IgG/total human IgG), in first-void urine from 63 women to monitor the immune response before and after vaccination with a prophylactic HPV vaccine (Gardasil9).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Prof, MD, PhD, Principal Investigator — Universiteit Antwerpen; Ilse De Coster, MD, Principal Investigator — Universiteit Antwerpen; Wiebren A. A. Tjalma, Prof, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- university of Antwerp - centre for the evaluation of vaccination, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No